CLINICAL TRIAL: NCT02172508
Title: A Randomised, Double-blind, Placebo-controlled 7-week Trial to Investigate the Effects of Tiotropium Inhalation Capsules (18 μg) Once Daily on Exercise Tolerance, Daily Activity and Dyspnoea in Patients With Chronic Obstructive Pulmonary Disease (COPD) Participating in 3 Weeks of Pulmonary Rehabilitation.
Brief Title: Effect of Tiotropium Inhalation Capsules on Exercise Tolerance, Daily Activity and Dyspnoea in Patients With Chronic Obstructive Pulmonary Disease (COPD) Participating in 3 Weeks of Pulmonary Rehabilitation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.289
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (2):
- Tiotropium (Experimental)
  Interventions: Drug: Tiotropium Inhalation Capsule
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Lactose Capsule

INTERVENTIONS:
Drug: Tiotropium Inhalation Capsule
  Arms: Tiotropium
Drug: Placebo Lactose Capsule
  Arms: Placebo

SUMMARY:
The primary objective of the study is to investigate the effect of the combined therapy 18 μg tiotropium q.d. plus pulmonary rehabilitation versus placebo plus pulmonary rehabilitation on 6-minute walking distance (6MWD) after 7 weeks of treatment in patients with moderate to severe COPD. The secondary objective of the study includes assessments of the effects of the combined therapy 18 μg Tiotropium q.d. plus rehabilitation versus placebo plus rehabilitation on dyspnoea, constant work rate exercise endurance, daily activity and lung volumes. The third objective of the study is to investigate the correlation between the results of the 6-minute walking test (6MWT), the constant work rate exercise test (CWR) and daily activity.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an Informed Consent Form consistent with ICH-GCP guidelines prior to participation in the trial, which might include pre-study washout of their usual pulmonary medications and restrictions.
2. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:

   Patients must have relatively stable airway obstruction with an FEV1 ≤ 65% of predicted normal and FEV1 ≤ 70% of FVC on visit 1 and 3.
3. Patients must show TGV ≥ 120% of predicted normal
4. Male or female patients ≥ 40 but ≤ 75 years old
5. Patients must be current or ex-smokers with a smoking history of more than 10 pack-years.
6. Patients must be able to perform all study related tests including the exercise tests, acceptable pulmonary function tests and must be able to maintain records during the study period as required in the protocol.
7. Patients must be able to inhale medication from the HandiHaler® and from a metered dose inhaler.
8. Patients must be already eligible for participation in a pulmonary rehabilitation program as per the investigator's usual criteria.

Exclusion Criteria:

1. Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease which, in the opinion of the investigator, may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
2. Patients with clinically relevant abnormal baseline hematology, blood chemistry or urinanalysis, if the abnormality defines a disease listed as an exclusion criterion.
3. All patients with an serum glutamic-oxaloacetic transaminase (SGOT) > 80 IU/L, serum glutamic-pyruvic transaminase (SGPT) > 80 IU/L, bilirubin > 2.0 mg/dL or creatinine > 2.0 mg/dL will be excluded regardless of clinical condition.
4. Patients with a history of asthma, allergic rhinitis or atopy or who have a total blood eosinophil count > 600/mm3. A repeat eosinophil count will not be conducted in these patients.
5. Patients with a recent history (i.e., six months or less) of myocardial infarction.
6. Patients with unstable or life-threatening cardiac arrhythmias, including any patient with a newly diagnosed, clinically relevant arrhythmia on the ECG performed on visit 1. Patients with arrhythmias requiring an intervention (i.e. hospitalization, cardioversion, pacemaker placement, and automatic implantable cardiac defibrillator (AICD) placement) or a change in drug therapy during the last year should also be excluded from the study.
7. Patients who have been hospitalized for heart failure during the past three years.
8. Patients with known active tuberculosis.
9. Patients with a history of cancer within the last 5 years. Patients with treated basal cell carcinoma are allowed.
10. Patients with a history of cystic fibrosis, bronchiectasis, interstitial lung disease, or pulmonary thromboembolic disease.
11. Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion 1.
12. Patients with any respiratory infection in the 4 weeks prior to the screening visit and recovery within 6 weeks prior to visit 3 should be randomised 6 weeks following recovery from the infection or exacerbation.
13. Patients who are currently in a pulmonary or cardiac rehabilitation program or who have completed a pulmonary or cardiac rehabilitation program in the last 6 months prior to the screening visit (visit 1).
14. Patients with known hypersensitivity to anticholinergic drugs, lactose or any other components of the inhalation capsule delivery system.
15. Patients with symptomatic prostatic hyperplasia or bladder neck obstruction. Patients being treated for prostatic hyperplasia and report minimal symptoms may be included and should continue their medications.
16. Patients with known narrow-angle glaucoma.
17. Patients with a theophylline level > 5.0 μg/ml.
18. Patients who are currently on β-blocker therapy including ocular preparations.
19. Patients who are being treated with oral beta-adrenergics.
20. Patients who are being treated with antihistamines (H1 receptor antagonists) for asthma or excluded allergic conditions (See exclusion criterion No. 4).
21. Patients using oral corticosteroid medication at unstable doses (i.e., less than 6 weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
22. Patients who are being treated with monamine oxidase inhibitors or tricyclic antidepressants.
23. Patients who have been treated with commercially available Spiriva® within the last 3 months prior to visit 1.
24. Patients who are being treated with cromolyn sodium or nedocromil sodium within 1 month of visit 1.
25. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception for the previous three months (i.e., oral contraceptives, intrauterine devices, diaphragm or subdermal implants e. g.: Norplant®).
26. Significant alcohol or drug abuse within the past 5 years.
27. Current participation in any other clinical trial or use of any investigational drug within one month or six half lives (whichever is greater) prior to screening visit (visit 1).
28. Patients who use supplemental oxygen while at rest should be excluded.
29. Patients with oxygen saturation below 85% during exercise despite supplemental oxygen therapy at visits 1 and 2 will be excluded from further participation.
30. If in the investigator's opinion patients can only perform exercise testing with supplemental oxygen, supplemental oxygen therapy will be used at all following tests including rehabilitation program under constant level.
31. Patients with a history of orthopedic, muscular or neurologic disease that would interfere with regular participation in aerobic exercise or with exercise testing.
32. Patients with a body mass index > 30 kg/m2 or < 18 kg/m2.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-01; Primary Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 6 Minute Walking Distance (6MWD) | Baseline, day 51

SECONDARY OUTCOMES:
Dyspnoea at the end of the 6MWT determined by the Modified Borg Scale (Dyspnoea Borg 6MWT), | Up to day 51
Endurance time during a constant work rate exercise test (CWR) | Up to day 51
Forced expiratory volume in one second (FEV1) | Up to day 51
Forced vital capacity (FVC) | Up to day 51
Slow vital capacity (SVC) | Up to day 51
Total lung capacity (TLC) | Up to day 51
COPD symptom scores (wheezing, shortness of breath, coughing, and tightness of chest) | Up to day 51
Transition Dyspnoea Indices (TDI) | Up to day 51
Change from baseline in Chronic Respiratory Questionnaire (CRQ), | Baseline, up to day 51
Change from baseline in patient's global evaluation on an 8-point-scale | Baseline, up to day 51
Amount of rescue medication used | Up to day 51
Daily physical activity, measured by a pedometer as number of registered activity impulses per day | Up to day 51
Total duration of endurance training on cycle ergometer during rehabilitation period | Up to day 51
Occurrence of adverse events | Up to day 51
Static Inspiratory capacity (IC) | Up to day 51
Residual volume (RV) | Up to day 51
Thoracic gas volume (TGV) | Up to day 51
Airways resistance (Raw) | Up to day 51
Change from baseline in blood pressure | Baseline, day 51
Change from baseline in pulse rate | Baseline, day 51
Change from baseline in laboratory tests | Baseline, day 51
Change from baseline in electrocardiogram (ECG) | Baseline, day 51
Change from baseline in physician's global evaluation on an 8-point-scale | Baseline, up to day 51